CLINICAL TRIAL: NCT03494959
Title: Pentaglobin As Early Adjuvant Treatment for Febrile Neutropenia in Acute Leukemia or Allogeneic Hematopoietic Stem Cell Transplant Patients Colonized by Carbapenem-resistant Enterobacteriaceae (CRE) or Pseudomonas Aeruginosa (PA)
Brief Title: Pentaglobin in CRE and PA Neutropenic Infections
Acronym: PENTALLO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GITMO PENTALLO; 2018-001344-57 (EudraCT Number)
Record Dates: First submitted 2018-04-05; First posted 2018-04-11 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Septic Shock
Keywords: Pentaglobin; Carbapenem-resistant Klebsiella pneumoniae; Pseudomonas aeruginosa; febrile neutropenia; infection-related mortality
MeSH Terms: conditions — Shock, Septic; Pseudomonas Infections; Febrile Neutropenia | interventions — pentaglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Pentaglobin (Experimental): Patients should receive the best available first-line therapy, usually a combination therapy, based on the in vitro susceptibility results of the pre-treatment screening swab in combination to Pentaglobin 5ml/kg over a 12h i.v. infusion for 3 consecutive days.
  Interventions: Drug: Pentaglobin

INTERVENTIONS:
Drug: Pentaglobin — Antimicrobial treatment active against the multidrug-resistant strain should be started in case of neutropenic fever (oral temperature ≥38.3°C or temperature ≥38.0°C sustained over a one-hour period). Patients should receive the best available first-line therapy, usually a combination therapy, based on the in vitro susceptibility results of the pre-treatment screening swab in combination to Pentaglobin 5ml/kg over a 12h i.v. infusion for 3 consecutive days. Empirical treatment should be subsequently streamlined according to microbiological results (both positive and negative). Pentaglobin should be started within 12h from the onset of fever, regardless of the presence of hemodynamic stability.

SUMMARY:
To demonstrate that the early addition of Pentaglobin to the best available antimicrobial therapy is able to reduce mortality and improve survival in neutropenic febrile acute leukemia or allo- Hematopoietic stem cell transplantation (HSCT) patients colonized by carbapenem-resistant Enterobacteriaceae or by any Pseudomonas aeruginosa.

DETAILED DESCRIPTION:
The study will enroll adult patients suffering from acute leukemia candidate to intensive chemotherapy or patients with hematological cancers candidate to allogeneic transplant with a documented colonization or previous bloodstream infection sustained by Carbapenem-resistant Enterobacteriaceae or Pseudomonas aeruginosa.

Primary objective: to demonstrate that the early addition of Pentaglobin to the best available antimicrobial therapy is able to reduce mortality and improve survival in neutropenic febrile acute leukemia or allo- Hematopoietic stem cell transplantation (HSCT) patients colonized by carbapenem-resistant Enterobacteriaceae or by any Pseudomonas aeruginosa.

Secondary Objectives: to evaluate the overall impact of Pentaglobin administration in the study population concerning infectious complications and treatment-related mortality.

This study will have two co-primary endpoints:

To demonstrate a 50% reduction in 30-day mortality for carriers developing a pre-engraftment bloodstream infection sustained by carbapenem-resistant Enterobacteriaceae or Pseudomonas aeruginosa (earlier primary endpoint).

To increase the Overall Survival (OS) at 4 months from the start of intensive treatment in all carriers of CRE or PA compared to historical controls (later primary endpoint)

Secondary endpoint are:

OS in carriers not developing a bloodstream infection sustained by carbapenem-resistant Enterobacteriaceae (CRE) or Pseudomonas aeruginosa (PA) at 4 months from the start of intensive chemotherapy or transplant Days of fever > 38.3°C within 4 months from the start of start of intensive chemotherapy or transplant Days of hospitalization within 4 months from the start of intensive chemotherapy or transplant Days of i.v. antimicrobials within 4 months from the start of intensive chemotherapy or transplant Non-relapse mortality (NRM) at 4 months from the start of intensive chemotherapy or transplant Patients will be treated according to the standard procedures, which will be decided by each Center according to local policies (e.g. chemotherapy cycles for acute leukemia, choice of conditioning regimen for allo- Hematopoietic stem cell transplantation and graft-versus-host- disease prophylaxis, anti-microbial prophylaxis).

Pre-treatment microbiological screening Before the initiation of intensive chemotherapy (within 2 weeks) patients will be screened by rectal and pharyngeal swabbing for multidrug-resistant Gram-negative bacilli, as part of routine clinical practice.

If the rectal and/or pharyngeal swabs reveal the presence of Carbapenem-resistant Enterobacteriaceae or Pseudomonas aeruginosa, the patient will be considered eligible for the study.

Patients with a previous documented infection (within 3 months) caused by Carbapenem-resistant Enterobacteriaceae or Pseudomonas aeruginosa are also considered eligible for the study regardless of the result of the rectal/pharyngeal swabs.

Treatment and management of febrile neutropenia in Carbapenem-resistant Enterobacteriaceae or Pseudomonas aeruginosa carriers Antimicrobial treatment active against the multidrug-resistant strain should be started in case of neutropenic fever, defined as a single oral temperature of ≥38.3°C or a temperature of ≥38.0°C sustained over a one-hour period.

At the onset of neutropenic fever and before the initiation of antimicrobial therapy at least 2 sets of blood cultures (2 bottles from a peripheral vein and 2 bottles from central venous catheter) should be performed.

Patients should receive the best available first-line therapy, usually a combination therapy, based on the in vitro susceptibility results of the pre-treatment screening swab in combination to Pentaglobin 5ml/kg over a 12h i.v. infusion for 3 consecutive days. Empirical treatment should be subsequently streamlined according to microbiological results (both positive and negative) Pentaglobin should be started within 12h from the onset of fever, regardless of the presence of hemodynamic stability.

Septic shock should be diagnosed and managed according to standard procedure The duration of the antimicrobial therapy or subsequent lines of therapy will be decided by local investigators according to clinical judgment. Cycles of Pentaglobin can be repeated according to clinician judgment (usually at least 1 week).

In this study two co-primary endpoints will be evaluated: the 30-day mortality rate for carriers developing a pre-engraftment bloodstream infection sustained by Carbapenem-resistant Enterobacteriaceae or Pseudomonas aeruginosa and the Overall Survival at 4 months from the start of intensive treatment in pre-treatment carriers.

In order to address the multiplicity issue, the Bonferroni method to adjust the significance level will be applied as follows:

* the early endpoint (i.e. the "30-day mortality for carriers developing a pre-engraftment bloodstream infection sustained by CRE or PA") will be tested at the 3.0% significance level using the Simon (minimax) phase II study design;
* the late endpoint (i.e. the "OS at 4 months from the start of intensive treatment in pre-treatment carriers") will be tested at the 2.0% significance level.

Adaptive study design

Early primary endpoint:

30-day mortality rate for carriers developing a pre-engraftment bloodstream infection sustained by Carbapenem-resistant Enterobacteriaceae or Pseudomonas aeruginosa.

The test was planned to determine whether it will be possible to obtain a consistent rate of reduction in 30-day mortality for carriers developing a pre-engraftment bloodstream infection sustained by CRE or PA. In the proposal, to reject the null hypothesis that p<=0.60 (mortality rate: 0.40) vs. the alternative hypothesis that p>=0.80 (mortality rate: 0.20) with Type I error probability (α) equal to 0.03 and 80% power (1-β), a maximum of 40 evaluable patients has to be accrued.

In the first stage of the study, 31 evaluable patients will be enrolled and the trial will be terminated if 9 or more patients died by day +30; otherwise, 9 further evaluable patients will be enrolled in the second stage.

If the total number of patients died will be less than or equal to 11, the combination therapy will not be recommended for further studies.

If the total number of patients alive at day +30 is at least 30, the treatment will be deemed worthy of further investigations.

Considering that approximately 33% of enrolled patients will be "carriers developing a pre-engraftment bloodstream infection sustained by CRE or PA", a total of 120 patients will be needed to be enrolled.

So, considering the study design, an interim analysis is planned after 31 carriers developing a pre-engraftment bloodstream infection sustained by CRE or PA.

Late primary endpoint:

Overall Survival at 4 months from the start of intensive treatment in pre-treatment Carbapenem-resistant Enterobacteriaceae or Pseudomonas aeruginosa carriers.

The later endpoint is the Overall Survival at 4 months. This sample size was calculated using the "Sample size tables for exact single-stage phase II design" (A'Hern RP, Statistics in Medicine 2001). Considering an expected Overall Survival at 4 months of 70% from the start of intensive treatment in pre-treatment carriers, the number of patients required to evaluate an increase on the Overall Survival from 50% (P0) to 70% (P1) with 90% power at the 2.0% significance level (one side) is 68.

So, the total number of patients to be enrolled in this study is 120, including the 68 patients needed for the later endpoint. Calculations were made using PASS software.

The Data Safety Monitoring Board will make one monitoring at 31 evaluable patients (in concomitant with the interim analysis) to ensure the safety of patients enrolled in to the study.

The end of enrollment will end based on the ad interim analysis results according to the adaptive model of the study.

Enrollment may then terminate after the interim analysis provided after recording 31 bacteremia in 31 patients with CRE or PA or when the 120th patient will be enrolled.

Each patient enrolled will have a minimum follow-up period of 4 months from transplant or start chemotherapy.

Each patient enrolled developing bacteremia sustained by Carbapenem-resistant Enterobacteriaceae or Pseudomonas aeruginosa will have a 30-day follow-up from initiation of treatment with Pentaglobin.

It is planned to complete the total enrollment (120 patients) in 2 years starting from the first patient enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* Performance status: ECOG <3
* Diagnosis of acute myeloid leukemia or acute lymphoblastic leukemia candidate to intensive chemotherapy
* Indication to allogeneic Hematopoietic stem cell transplantation (HSCT) for hematological cancers, including severe aplastic anemia (second transplants allowed)
* Pre-treatment colonization by Carbapenem-resistant Enterobacteriaceae (CRE) or Pseudomonas aeruginosa (PA) documented by rectal and/or pharyngeal swab.
* Pre-treatment bloodstream infection sustained by CRE or PA.
* Written and signed informed consent

Exclusion Criteria:

* Uncontrolled systemic infection
* Anaphylaxis or severe prior reactions to immunoglobulins preparation
* Severe concomitant illness:

  * patients with severe renal impairment, i.e. patients on dialysis or prior renal transplantation or S-creatinine > 3.0 x ULN or calculated (CKD-EPI) creatinine-clearance < 50 ml/min
  * patients with severe pulmonary impairment (DLCOSB (Hb-adjusted)/or FEV1 < 50 % or severe dyspnea at rest or requiring oxygen supply);
  * patients with severe cardiac impairment (LVEF < 40 %)
  * patients with severe hepatic impairment (hyperbilirubinemia > 3 x ULN or ALT / AST > 5 x ULN).
* patients who on the basis of the investigator's consideration are not able to give the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-12-06 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Sepsis-related mortality | day +30 from the onset of neutropenic fever
  Sepsis-related mortality is considered as the time from the onset of neutropenic fever to death caused by uncontrolled documented infection, in the absence of any other interfering cause of death
Overall Survival | at 4 months from the start of intensive treatment
  is defined as the probability of survival irrespective of disease state at any point in time. Patients alive at their last follow-up are censored. It is analyzed by the Kaplan-Meier method, Log-Rank Test and parametric or semiparametric survival models.
Non-Relapse Mortality | at 4 months from the start of intensive treatment.
  It is defined as the probability of dying without previous occurrence of a relapse, which is a competing event

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Ciceri, Principal Investigator — Ospedale San Rafafele
Locations (20):
- Italy (20):
  - Ospedale Binaghi, Cagliari, Italy
  - Ospedale Cardarelli, Napoli, napoli
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti, Ancona
  - Policlinico di Bari-Ematologia con trapianti, Bari
  - Ospedale San Orsola, Bologna
  - AO Spedali Civili di Brescia- USD - TMO Adulti, Brescia
  - S.C. Ematologia - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Cattedra di Ematologia - Azienda Ospedaliera di Careggi, Florence
  - Ematologia e Centro Trapianti Midollo Osseo - Ospedale IRCCS Casa Sollievo della Sofferenza, Foggia
  - Trapianti Midollo Osseo - Policlinico S. Martino, Genova
  - Policlinico VIto Fazzi, Lecce
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Ospedale G. Da Saliceto di Piacenza, Piacenza
  - Cattedra di Ematologia - Policlinico, Roma
  - Divisione di Ematologia - Istituto di Semeiotica Medica - Policlinico A. Gemelli, Roma
  - Policlinico Universitario Tor Vergata, Roma
  - Ospedale Moscati, Taranto
  - AOU CIttà della Salute e della Scienza, Torino
  - Clinica Ematologica - Policlinico Universitario, Udine

IPD SHARING:
Plan to Share IPD: No